CLINICAL TRIAL: NCT02930577
Title: Factors Associated With Treatment Adherence in Substance Users
Brief Title: Treatment Adherence in Substance Users
Acronym: TASU
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TOX-2015-71
Record Dates: First submitted 2016-08-26; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Substance-Related Disorders
Keywords: treatment adherence; outpatient treatment; drug dependence
MeSH Terms: conditions — Substance-Related Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Patients who completed addiction treatment between November 2013 and January 2016
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study evaluates the factors associated with treatment adherence in substance users. Differences in the level of adherence to treatment according to patient-related factors, addiction and treatment are analyzed. The individual effect of each factor on treatment adherence is assessed.

DETAILED DESCRIPTION:
INTRODUCTION: Treatment dropout is an unsolved problem in the addiction process which makes frequent the failure of the addiction therapy. Research shows that the majority of dropouts occur during the first weeks of the treatment. These are the most serious ones because they have the worst prognosis. Some factors, related to the patients and the therapy, have been associated with treatment dropout but the diversity of studied variables, the heterogeneity of patients and the sparse population of many studies, hampers external validity and comparison of results.

OBJECTIVES: Analyze the treatment adherence of an outpatient treatment program for addicts. Identify factors associated with treatment adherence in substance users.

MATERIAL AND METHODS: Observational, analytical, longitudinal and retrospective study in substance users who completed addiction treatment between November 2013 and January 2016. Treatment adherence is measured in terms of medical discharge, regular attendance at activities and success in the NOC indicators. Differences in the level of adherence to treatment according to patient-related factors, addiction and treatment are analyzed. The individual effect of each factor on treatment adherence is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Substance-Related Disorders
* Treatment for drug dependency

Exclusion Criteria:

* Admission for detoxification treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Substance users who completed addiction treatment between November 2013 and January 2016.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
treatment adherence | two month
  Good adherence: if the patient complete the treatment, attends health professionals sessions and/or gets a sufficient score in objectives nursing.
  Bad-adherence: if the patient not complete the treatment.

SECONDARY OUTCOMES:
gender | two months
  options: male or female.
age | two months
work situation | two months
  options: unemployed, worker, pensioner or student.
cohabitation | two months
  options: alone, with parents or with the couple and sons
family support | two months
  options: no support, support, support and groups
all mental disorders of DSM-IV (Diagnostic and Statistical Manual of mental Disorders) | two months
all drugs | two months
Self-esteem level according to the Rosenberg Self-Esteem questionnaire. | two months
  options: high, medium or low self-esteem level.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] López Goñi JJ, Fernández-Montalvo J, Arteaga A. El abandono (dropout) en el Tratamiento de la Adicción: Explorando las Características de los Pacientes. Am J Addict. 2011;(21):78-85.
- [Background] Zamora YR. Predicción del abandono del tratamiento en adictos mediante el cuestionario VPA-30. Revista del Hospital Psiquiátrico de La Habana. 2014;11(2).
- [Background] Sanchez-Hervas E, Secades-Villa R, Gomez FJ, Romaguera FZ, Garcia-Rodriguez O, Yanez EM, Frances MC, Fernandez GG. [Treatment dropout in cocaine addicts]. Adicciones. 2010;22(1):59-64. Spanish. PMID 20300715
- [Background] Valero-Aguayo L, Ortiz-Tallo M, Parra-García MM, Jiménez-Guerra M. Valoración de resultados y perfil psicosocial de un programa de rehabilitación de personas con drogodependencias. Anales de Psicología. 2013;29(1):38-47.
- [Background] Fernández-Montalvo J, López Goñi JJ, Landa N, Illescas C, Lorea, I, Zarzuela, A. Trastornos de personalidad y abandonos terapéuticos en pacientes adictos: resultados en una comunidad terapéutica. Int J Clin Health Psychol. 2004; 4(2): 271-283.
- [Background] Llinares Pellicer MC, Palau Munoz C, Albiach Catala C, Santos Diez P. [Predictive variables of adherence to treatment in alcoholics]. Actas Esp Psiquiatr. 2002 Nov-Dec;30(6):370-5. Spanish. PMID 12487947
- [Background] Garcia-Rodriguez O, Secades-Villa R, Alvarez Rodriguez H, Rio Rodriguez A, Fernandez-Hermida JR, Carballo JL, Errasti Perez JM, Al-Halabi Diaz S. [Effect of incentives on retention in an outpatient treatment for cocaine addicts]. Psicothema. 2007 Feb;19(1):134-9. Spanish. PMID 17295995
- [Background] Albiach C, Llinares MC, Palau C, Santos P. Adherencia en heroinómanos: la potencia predictiva de los estadios de cambio evaluados durante la admisión al tratamiento. Adicciones. 2000;12(2):225-234.
- [Background] Olmos-Espinosa R, Madoz-Gúrpide A, Ochoa E. Situación al año de los adictos a opiáceos que siguieron tratamiento ambulatorio tras desintoxicación hospitalaria. Adicciones. 2001;13(2):173-8.
- [Background] Albiach C, Palau C, Llinares C, Santos P. Estudio sobre la adherencia al tratamiento en sujetos con adicción a diferentes sustancias que acuden a servicios ambulatorios. En: V Encuentro Nacional sobre drogodependencias y su enfoque comunitario; 1998; Chiclana de la Frontera, Cádiz, p. 57-70.
- [Background] Herrera JM, Barberán M, Yumar T. La adherencia al tratamiento en una Unidad de Atención a las Drogodependencias (UAD). Trabajo Social y Salud. 2008; (61):155-182.
- [Background] López-Goñi JJ, Fernández-Montalvo J, Illescas C, Landa N, Lorea I. Razones para el abandono del tratamiento en una comunidad terapéutica. Trastor Adict. 2008;10(2):104-111.
- [Background] Domínguez-Martín AL, Miranda-Estribí MD, Pedrero-Pérez EJ, Pérez-López M, Puerta-García C. Estudio de las causas de abandono del tratamiento en un centro de atención a drogodependientes. Trastor Adict. 2008;10(2):112-120.
- [Background] Silva Lento AF, Cerqueira AM, Rocha Costa OC. Programa de deshabituación. ¿Cuáles son los factores que llevan al dropout? Revista española de drogodependencias. 2004; (1):62-70.
- [Background] Roncero C, Rodriguez-Cintas L, Barral C, Fuste G, Daigre C, Ramos-Quiroga JA, Casas M. Treatment adherence to treatment in substance users referred from Psychiatric Emergency service to outpatient treatment. Actas Esp Psiquiatr. 2012 Mar-Apr;40(2):63-9. Epub 2012 Mar 1. PMID 22508071
- [Background] Sirvent C, Villa M, Blanco P, Rivas C, Linares MP, Quintana L. Predicción del abandono (vs. éxito) terapéutico en adicciones. (Presentación del cuestionario VPA-30 (c Sirvent, 2009), de variables predictores de abandono y adherencia al tratamiento en adicciones). Interpsiquis 2010.
- [Background] Martinez-Gonzalez JM, Albein-Urios N, Verdejo-Garcia A, Lozano-Rojas O. [Differential aspects of treatment dropout risk in cocaine dependent patients with and without personality disorders]. Adicciones. 2014;26(2):116-25. Spanish. PMID 25288259
- [Background] Roncero C, Gomez-Baeza S, Vazquez JM, Teran A, Szerman N, Casas M, Bobes J. Perception of Spanish professionals on therapeutic adherence of dual diagnosis patients. Actas Esp Psiquiatr. 2013 Nov-Dec;41(6):319-29. Epub 2013 Nov 1. PMID 24203504
- See also: Presentación del cuestionario VPA-30 (c Sirvent, 2009), de variables predictores de abandono y adherencia al tratamiento en adicciones — http://www.researchgate.net/publication/271511182_Prediccin_del_abandono_(versus_xito)_teraputico_en_adicciones_Predict_the_therapeutic_abandon_(or_overcoming)_in_addictions
- See also: Resumen ejecutivo: Informe mundial sobre las drogas. Oficina de las Naciones Unidas contra la Droga y el Delito (UNODC); 2014. — http://www.unodc.org/documents/wdr2014/V1403603_spanish.pdf